CLINICAL TRIAL: NCT01778842
Title: PhaRmacodynamic Effect of Antiplatelet Agents in Elderly Patients: Standard Clopidogrel Versus prasugrEl Low Dose Therapy.
Brief Title: Standard Clopidogrel Versus Prasugrel Low Dose Therapy in Elderly Patients With Acute Coronary Syndrome
Acronym: RESET ELDERLY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESET ELDERLY
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
Keywords: antiplatelet effect; prasugrel; clopidogrel; acute coronary syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel low dose (Experimental): Patient will be randomized to this intervention will receive prasugrel 5 mg and after 15 days and 30 days we will control the responsivness of the study drug.
  Interventions: Drug: Prasugrel
- Clopidogrel standard dose (Experimental): Patient will be randomized to this intervention will receive clopidogrel 75 mg and after 15 days and 30 days we will control the responsivness of the study drug.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Patient will be randomized to this intervention will receive the standard dose of clopidogrel and after 15 days and 30 days we will control the responsivness of the study drug.
  Arms: Clopidogrel standard dose
Drug: Prasugrel — Patient will be randomized to this intervention will receive the low dose of prasugrel and after 15 days and 30 days we will control the responsivness of the study drug.
  Arms: Prasugrel low dose

SUMMARY:
The elderly represent a growing segment of the coronary population treated by dual antiplatelet therapy for percutaneous coronary intervention (PCI). These patients bear a higher risk of both ischemic events and bleeding complications than younger patients, with a subsequently higher rate of mortality.Recentprogress in antithrombotic treatment demonstrated the efficacy of adding a P2Y12 receptor antagonist to low-dose aspirin. Whether this benefit is also present in the elderly remains a debated issue due to the lack of specific data in this sub-population. The present study was realized to provide specific data on platelet response to clopidogrel, standard dose (75 mg) or prasugrel 5 mg in elderly patients (≥75 years old) whereas the superiority in PR response of the latter should allows the Prasugrel therapy in elderly patients with the better clinical efficacy and therapeutical safety already showed compared with Clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* PCI with stent implantation
* clopidogrel responsiveness
* > 75 years of age.

Exclusion Criteria:

* history of bleeding diathesis
* chronic oral anticoagulation treatment
* contraindications to antiplatelet therapy
* PCI or coronary artery bypass grafting (CABG) < 3 months
* hemodynamic instability
* platelet count < 100,000/μl
* hematocrit < 30%
* creatinine clearance < 25 ml/min
* Patients with a history of stroke
* other contraindication for prasugrel administration
* patients weighing < 60 kg
* high on treatment platelet reactivity

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
superiority of prasugrel low dose | 30 days
  The primary aim will be to investigate the antiplatelet effect of half dose of prasugrel (5 mg) versus standard dose of clopidogrel in patients with acute coronary syndrome and coronary diseases, treated with percutaneous coronary intervention and stent implantation.

SECONDARY OUTCOMES:
Bleeding | 12 months
  Bleeding (major, minor, or minimal according to the TIMI study criteria)
major adverse cardiac events | 12 months
  major adverse cardiac events (cardiovascular death, myocardial infarction, and stroke) will be evaluated during the all period of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Rome, Italy